CLINICAL TRIAL: NCT01706861
Title: A Post Market Study Evaluating the Safety, Device Perfomance and Possible Emergent Risks of Celotres in Preventing Recurrence in Keloid LEsions Treated Adjunctive to suRgical Excision. PMCS: EURO-KLEAR
Brief Title: A Post Market Study Evaluating the Safety, Device Perfomance and Possible Emergent Risks of Celotres in Preventing Recurrence in Keloid Lesions Treated Adjunctive to Surgical Excision
Acronym: EURO KLEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halscion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAL-302
Record Dates: First submitted 2012-10-03; First posted 2012-10-15 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-02

CONDITIONS: Earlobe Keloids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Celotres (Other): Celotres following surgical removal of earlobe keloid.
  Interventions: Device: Celotres

INTERVENTIONS:
Device: Celotres — Celotres following surgical removal of earlobe keloid.

SUMMARY:
The objective of the study is to actively gather additional information on safety, device performance and possible emergent risks following the use of Celotres in a post-market setting when used to reduce the recurrence rate, volume, appearance and/or symptoms associated with keloid scarring in subjects undergoing surgical excision of keloids as compared to the scientific literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients electing to undergo keloid excision procedure
* Patients able and willing to give written informed consent

Exclusion Criteria:

* Patients with a known or potential risk of allergy or sensitivity to products or substances containing porcine gelatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The incidence of device related adverse events | Assessed at treatment, suture removal, Months 1, 3, 6, 9 and 12
  Device safety is defined as the incidence of device related adverse events.
Recurrence of keloid post scar excision | Assessed at 1, 3, 6, 9 and 12 months
  Proportion of subjects with recurrence of keloid scar post excision defined as the presence of scar tissue volume >0.3cc

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | Assessed at Pre-treatment, Months 1, 3, 6, 9 and 12
Subject Dermatology Life Quality Index (DLQI) | Assessed at Pre-treatment, Months 1, 3, 6, 9 and 12
Device Performance Evaluation | Assessed at Day 1
  Questions related to packaging integrity and successful administration of product as assessed by the Principal Investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Bella, MD, Principal Investigator — The Westbourne Centre
Locations (6):
- Poland (4):
  - Angelius Szpital Proviat, Katowice
  - Oddzial Leczenia Oparzen Chirugil Plastysznej, Krakow
  - Kosmetyczno-Lekarska Spółdzielnia Pracy "IZIS", Warsaw
  - Wojskowy Oddzial Kliniczny ChirurgiiPlastycznej, Warsaw
- University of the West Indies, Nassau, The Bahamas
- The Westbourne Centre, Edgbaston, Birmingham, United Kingdom